CLINICAL TRIAL: NCT05736133
Title: Determining the Impact of a New Physiotherapist-Led Primary Care Model for Hip and Knee Pain - A Pilot Cluster Randomized Controlled Trial
Brief Title: Determining the Impact of a Physiotherapist-Led Primary Care Model for Hip and Knee Pain - A Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Miller, PT, PhD (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other)
Responsible Party: Sponsor-Investigator, Jordan Miller, PT, PhD, Assistant Professor, School of Rehabilitation Therapy, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6038205
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Papaverine

STUDY DESIGN:
Intervention Model Description: This is a pilot cluster randomized controlled trial randomizing 14 sites to the PT-led primary care model for hip/knee pain or to the usual care model
Masking Description: Due to the nature of the new model of care and comparison, it is not possible to blind the patient participants or health care providers. Since the primary outcomes are self-reported outcome measures, the assessor is also not blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led primary care model for hip and knee pain (Experimental): The index intervention will incorporate a PT within the primary care team and make them available at the first point of contact for people with hip or knee pain. There will be 4 key components of this intervention: 1) Initial assessment and screening; 2) Brief individualized intervention at first visit; 3) Health services navigation; 4) Providing additional PT care for people with an unmet need (e.g., no insurance coverage for PT).
  Interventions: Other: Physiotherapist-led primary care model for hip and knee pain
- Usual physician-led primary care model for hip and knee pain (Active Comparator): Participants will be seen by a primary care physician or a nurse practitioner, depending on the current practice at the clinic. Participants in both groups will be permitted to seek additional care outside of the primary care clinic.
  Interventions: Other: Usual physician-led primary care model for hip and knee pain

INTERVENTIONS:
Other: Physiotherapist-led primary care model for hip and knee pain — 1. Initial assessment and screening: The PT will provide a comprehensive assessment according to established clinical practice guidelines.
  2. Brief individualized intervention at first visit: The PT intervention will be at the discretion of the PT to reflect real-world PT intervention.
  3. Health services navigation: Participants will be provided with options available to them in their community for rehabilitation. For example, they may be referred to community PT for ongoing management or presented with group exercise options. Participants will be assessed regarding the need for specialist referrals or resources available to manage complex clinical presentations such as comorbidity or frailty. Participants may be referred to the primary care provider if no specialized services are needed or when the PT cannot provide a direct referral. All individuals may have their medications reviewed by a physician if deemed appropriate by the PT or requested by the participant.
  Arms: Physiotherapist-led primary care model for hip and knee pain
Other: Usual physician-led primary care model for hip and knee pain — The physician led primary care intervention will be unstandardized to best reflect standard clinical practice in Canada.
  Arms: Usual physician-led primary care model for hip and knee pain

SUMMARY:
This is a pilot cluster randomized controlled trial to to evaluate the individual and health system impacts of implementing a new physiotherapist-led primary care model for hip and knee pain in Canada.

DETAILED DESCRIPTION:
Arthritis is one of the leading causes of pain, disability, and reduced quality of life in patients. Arthritis currently affects one in five Canadians (six million), which is expected to rise to nine million people by 2040. Osteoarthritis (OA) is the most common forms of arthritis, with hip and knee being two of the most common locations.

For most people, the first point of contact for their pain is their primary care provider. Due to the rise in patients seeking support at the primary care level, the shortage of primary care providers, and the high burden on these providers, patients often do not receive timely access to the care they require. A promising strategy is to have an integrated model of care where a physiotherapist (PT) is the first point of contact within interprofessional primary care teams. PTs can provide a comprehensive and efficient management strategy for patients presenting to their primary care provider with hip and knee pain complaints.

This study aims to determine the feasibility of conducting a cluster randomized trial in primary care settings in Ontario to evaluate the individual health outcomes and health system impact of implementing a new physiotherapist-led primary care model for people with hip and knee pain.

The primary objectives of this pilot study are:

1. Determine the feasibility of participant recruitment, assessment procedures, and retention.
2. Determine the feasibility of implementing a new PT led primary care model for hip and knee pain.
3. Explore the perspectives of patient participants and HCPs related to their experiences and attitudes towards the new service delivery model, barriers/facilitators to implementation, perceived satisfaction, perceived value and impact on clinic processes and patient participant outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Adults >= 19 years who ask to book a primary care visits where the primary reason is for hip or knee pain of any duration.

Exclusion Criteria:

* Cannot understand, read, and write English
* Known cancer causing hip or knee pain

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Participant Recruitment Rate | 20 weeks
  A full trial will be feasible if the investigators are able to recruit 1.5 participants per week per site over 20 weeks
Assessment Procedures | 12 months
  The investigators consider ≥80% of all assessment items completed and a mean time for completion of ≤60 minutes acceptable.
Retention | 12 months
  The investigators consider an attrition rate of ≤20% at 12-month follow-up successful. ≤35% attrition will be considered partially successful; however, additional retention strategies would be required for the full trial based on evidence that ≥20% attrition threatens trial validity
PT Treatment Fidelity | 20 weeks
  Treatment fidelity will be measured through an audit of a PT fidelity checklist and electronic medical record (EMR) to determine the consistency of the care provided. An acceptable level of fidelity will be considered ≥80% for each intervention component.

SECONDARY OUTCOMES:
Self-Reported Functioning | Baseline and 3, 6, 9, and 12 months follow-up
  Self-report using the Lower Extremity Functional Scale (0-80 score with higher score representing higher function)
Self-Reported Pain Intensity | Baseline and 3, 6, 9, and 12 months follow-up
  Measured using a numeric pain rating scale from 0 to 10 with higher scores indicating greater pain intensity.
Health-Related Quality of Life | Baseline and 3, 6, 9, and 12 months follow-up
  Measured using the EuroQoL-5D-5L (0 to 100 with greater scores indicating greater self-reported health related quality of life)
Pain Self Efficacy | Baseline and 3, 6, 9, and 12 months follow-up
  Confidence in abilities to participate in usual activities using the Pain Self Efficacy Questionnaire
Catastrophic Thinking | Baseline and 3, 6, 9, and 12 months follow-up
  Measured using the Pain Catastrophizing Scale (0 to 52 with higher scores indicating greater catastrophic thinking)
Fear of Movement | Baseline and 3, 6, 9, and 12 months follow-up
  Measured using the Tampa Scale of Kinesiophobia (an 11-item questionnaire)
Depression Subscale | Baseline and 3, 6, 9, and 12 months follow-up
  Measured using the 2-Item Patient Health Questionnaire
Global Rating of Change | 3, 6, 9, and 12 months follow-up
  Measured using an 11-point scale (-5 to +5 with negative scores indicating a worsening of physical functioning and positive scores indicating an improvement of physical functioning)
Satisfaction with Health Care | 3, 6, 9, and 12 months follow-up
  Measured using an 11-point scale(-5 to +5 with negative scores indicating a dissatisfaction with health care received and positive scores indicating satisfaction with health care received)
Adverse Events | 3, 6, 9, and 12 months follow-up
  Measured using an adverse events questionnaire that asks 1) if the participant has experienced any adverse events as a result of the treatments received (yes/no); 2) how long the event lasted (hours or days); 3) how severe the adverse event was (0-10 scale); 4) what adverse events were experienced.
Health Care Accessibility | Baseline
  Percentage of participants assessed within 48 hours of calling for an appointment
Health-Care Utilization - Consultations in Electronic Medical Record (EMR) | 12 months
  Number of consultations with primary care team members for hip or knee pain (e.g., physicians, nurse practitioners, nurses, social workers, occupational therapists)
Health-Care Utilization Survey - Visits to health professionals | 12 months
  Survey questions related to hip or knee pain: number of visits to health professionals outside the primary care team (e.g., chiropractors, massage therapists, occupational therapists, physiotherapists, chronic pain clinics)
Health-Care Utilization Survey - Medications | 12 months
  Survey questions related to hip or knee pain: number of medications taken. Includes type of medication, dose, frequency
Health-Care Utilization Survey - Walk-In Clinic Visits | 12 months
  Survey questions related to hip or knee pain: number of walk-in clinic visits outside of primary care centre
Health-Care Utilization Survey - Emergency Department Visits | 12 months
  Survey questions related to hip or knee pain: number of emergency department visits
Health-Care Utilization Survey - Inpatient Hospital Stays | 12 months
  Survey questions related to hip or knee pain: number of overnight hospital stays
Health-Care Utilization Survey - Surgeries, Procedures, Injections | 12 months
  Survey questions related to hip or knee pain: number of surgeries, procedures, and injections
Health-Care Utilization Survey - Specialist Visits | 12 months
  Survey questions related to hip or knee pain: number of visits to specialists
Health-Care Utilization Survey - Diagnostic Imaging | 12 months
  Survey questions related to hip or knee pain: number of diagnostic images received
Process Outcome - Medications Prescibed | 12 months
  Collected from the EMR: medications prescribed for hip or knee pain. Includes the type of medication prescribed
Process Outcome - Diagnostic Imaging Ordered | 12 months
  Collected from the EMR: diagnostic images ordered for hip or knee pain
Process Outcome - Exercises Prescribed | 12 months
  Collected from the EMR: exercises prescribed for hip or knee pain
Process Outcome - Education Provided | 12 months
  Collected from the EMR: education provided for hip or knee pain
Process Outcome - Referrals to other health care providers (HCPs) | 12 months
  Collected from the EMR: referrals to other HCPs (both internal and external to the primary health care team) for hip or knee pain
Process Outcome - Primary Care Visits | 12 months
  Collected from the EMR: visits to the primary care team for hip or knee pain
Process Outcome - Notes to Employers or Insurers | 12 months
  Collected from the EMR: notes provided to employers or insurers for hip or knee pain
Self-Report Time Lost | 12 months
  Self-reported time lost from work, volunteering, homemaking, and educational activities
Assistance Needed | 12 months
  Self-reported assistance needed, due to hip or knee pain, for self-care, housework, shopping, or transportation
Extra Expenses | 12 months
  Any extra expenses incurred as a result of hip or knee pain. Self-report
Cost Outcomes | 12 months
  Costs associated with all health utilization, self-reported time lost, assistance needed, and extra expenses. Will be presented as aggregate and time-specific costs

OTHER OUTCOMES:
Baseline Characteristics | Baseline
  To describe the study population, the investigators will capture the following through the survey: age, sex, gender, duration of musculoskeletal pain, locations of pain, medications, comorbidities, current work status, income, rurality, and ethnicity.
Comorbidities | Baseline
  Measured at baseline using the Functional Comorbidity Index (an 18-item list of comorbidities that are associated with physical functioning).
Chronicity of Pain | Baseline
  Self-reported length of time since current and first incidence of hip or knee pain
Participant Treatment Fidelity | 3 months follow-up
  Self-report adherence to PT advice

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The is no plan to share individual IPD with other researchers